CLINICAL TRIAL: NCT04645719
Title: Best Dose of Magnesium Sulfate Infusion in Obese. A Blind and Randomized Trial
Brief Title: Dose of Magnesium Sulfate Infusion in Obese
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 33298720.0.0000.5448
Record Dates: First submitted 2020-11-16; First posted 2020-11-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Obese; Analgesia
MeSH Terms: conditions — Obesity; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized and covered clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A professional will arrange the electronic draw, allocate the groups and prepare the opaque envelopes. Another professional will prepare the covert solution, the prescription of which will be inside the opaque envelope. The third professional will administer the anesthesia. Another team member will collect the data and organize it in a spreadsheet. The data will be analyzed by an independent statistician. Participants and performers for each stage will be covered for each participant's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactate ringer group (Placebo Comparator): Patients will receive only general anesthesia
  Interventions: Other: Lactate ringer group
- Real weight group (Active Comparator): Patients who will receive general anesthesia and magnesium sulfate infused at a dose of 15 mg.kg-1.h-1 based on the actual body weight
  Interventions: Drug: Magnesium sulfate dose through real weight group
- Corrected ideal weight group (Active Comparator): Patients who will receive general anesthesia and magnesium sulfate infused at a dose of 15 mg.kg-1.h-1 based on the corrected ideal weight
  Interventions: Drug: Magnesium sulfate dose through corrected ideal weight group

INTERVENTIONS:
Other: Lactate ringer group — General anesthesia only
  Other Names: Placebo comparator
  Arms: Lactate ringer group
Drug: Magnesium sulfate dose through real weight group — General anesthesia + magnesium sulfate 15 mg.kg-1.h-1 based on the patient's real weight
  Other Names: Active comparator 1
  Arms: Real weight group
Drug: Magnesium sulfate dose through corrected ideal weight group — General anesthesia + magnesium sulfate 15 mg.kg-1.h-1 based on the patient's corrected ideal weight
  Other Names: Active comparator 2
  Arms: Corrected ideal weight group

SUMMARY:
Magnesium sulfate has been shown to be a successful tool in a large number of clinical areas. Its benefits include neuroprotection, control of eclampsia / pre-eclampsia, control of intraoperative blood pressure, decreased neuroendocrine response during laryngoscopy and tracheal intubation and reduced levels of postoperative pain and consumption of analgesic.

Obese patients have become more and more frequent in the operating rooms, due to the increasing prevalence of this population worldwide. However, although they have received magnesium sulfate as part of the analgesic strategy in many centers, there has been no study demonstrating the appropriate dose of this medication in obese patients.

This study aims to compare two doses of magnesium sulfate in obese patients: based on their real weight or based on ideal weight.

DETAILED DESCRIPTION:
After approval by the Research Ethics Committee and registration of the project at ClinicalTrials (www.ClinicalTrials.gov) 75 patients will be selected from a population of obese patients scheduled for laparoscopic, bariatric or cholecystectomy surgery, who voluntarily accept to participate in the study. These participants will be distributed through an electronic draw in three groups. In the lactate ringer group (LRG), patients who will receive only general anesthesia will be grouped. In the real weight group (RWG) will be the patients who will receive general anesthesia and magnesium sulfate infused at a dose of 15 mg.kg-1.h-1 based on the actual body weight. In the corrected ideal weight group (CWG) will be the patients who will receive general anesthesia and the same dose of magnesium sulfate, but based on the corrected ideal weigh.

Inclusion criteria: patients aged 18 to 60 years, status I or II of the American Society of Anesthesiology, body mass index> 30 kg.m-2, scheduled for laparoscopic, bariatric surgery or cholecystectomy. Patients with allergies to any of the components of the protocol, who refuse to participate or sign the consent form, presenting neuromuscular impairment, heart block greater than first-degree atrioventricular block, using illicit drugs, with neuropsychiatric impairment, in blockers calcium channels and with renal impairment will not be invited to participate in the study.

A pre-trial phase will include 10 patients with a body mass index between 20 and 30 kg / m². These patients will receive magnesium sulfate infusion at a dose of 15 mg.kg-1h-1, and serial samples will be collected (before administration, 15, 30, 60, 120 and 240 min after administration) for comparison with the trial patients.

For this study, the sample size was determined to a level of 95% confidence, power equal to 80% and effect size of 0.40, a sample of 22 individuals was calculated for each of the 3 groups, adding a total of 66 participants. We rounded up to 25 participants per group to compensate for losses, with a total of 75 participants.

The result of the group draw will be kept hidden for participants and the team. Each participant will have an opaque envelope with their name and number corresponding to the order of entry into the study. The group each patient belongs to and the medication to be administered according to the group will be described on an identification card inside the envelope. A team member will be responsible for opening the envelope and preparing the medication to be administered, keeping the secret to the other study participants.

Participants will not receive pre-anesthetic medication. Upon arriving at the operating room, they will be monitored with continuous electrocardioscope, pulse oximetry, non-invasive blood pressure and monitoring of the level of consciousness. When the venous catheter is installed, the first blood sample (2 ml) will be collected to measure blood magnesium concentration. After blood collection, an infusion of the study comparison solution will be started as described below.

LRG - Ringer with lactate 16 ml.h-1 RWG - magnesium sulfate 15 mg.kg-1.h-1 based on the patient's real weight CWG - magnesium sulfate 15 mg / kg / h based on the patient's corrected ideal weight.

A professional will be assigned to prepare the syringe and pump to administer the substance in a covered manner to the patient and other team members. The infusion will be stopped at the end of the surgery. The professional who deals with the pump and substance corresponding to the patient's group will not participate in another stage of the study.

At the time of induction, all participants in the 3 groups will receive dipyrone 10 mg.kg-1, clonidine 2 µg.kg-1, cefazolin 2 g, dexamethasone 4 mg, ketoprofen 100 mg, ranitidine 50 mg, lidocaine 1.5 mg.kg-1. Pre-oxygenation with inspired fraction of 100% oxygen will be initiated for 3 min, followed by propofol in target-controlled infusion (TCI - target controlled infusion) with initial target at 4 µg.ml-1 (pharmacokinetic model Marsh, with target effect) guided by the monitoring of anesthetic depth. At that moment, the muscle relaxation monitor (TOF - train of four) will be calibrated, followed by the administration of 0.1 mg of cisatracurium and the start of remifentanil infusion in TCI to an effect concentration of 5 ng.ml-1. Anesthesia maintenance will be based on propofol in TCI guided by anesthetic depth monitoring, remifentanil (target 3 to 5 ng.ml-1) and cisatracurium 0.03 mg.kg-1 if TOF ≥ 2. There will be no additional dose of cisatracurium in the last 20 minutes surgery, unless necessary by the surgeon. The infusion of remifentanil will be controlled to prevent systolic blood pressure from reaching values greater than or less than 30% of baseline values, or a maximum of 130 mmHg and a minimum of 90 mmHg. At the end of surgery, after TOF> 2, patients will receive atropine 20 µg.kg-1 and neostigmine 40 µg.kg-1. Blood will be collected to examine the blood concentration of magnesium in all patients in the 3 groups at the time of venipuncture and 15, 30, 60, 120 and 240 min after the beginning of the covered solution.

Before extubation, all patients will receive an intravenous dose of morphine 0.05 mg.kg-1 and dipyrone 10 mg.kg-1. Five minutes after extubation, and then every 30 min, this dose of morphine will be repeated in case of pain greater than 3 on the verbal pain scale (scale from 0 to 10).

The following will be recorded and analyzed:

1. Blood concentrations of magnesium at the moments described
2. Consumption of painkillers upon awakening and during hospital stay
3. Cisatracurium latency (from injection to TOF = 0)
4. Cisatracurium duration 25 (from injection to TOF = 25%)
5. Total duration of cisatracurium (from injection to TOF = 90%)
6. Cisatracurium recovery index (between TOF 25% and 75%)

ELIGIBILITY:
Inclusion Criteria: healthy patients, patients with controlled systemic disease (arterial hypertension, endocrine disease), obese patients.

-

Exclusion Criteria: heart block, illicit drugs use, with neuropsychiatric impairment, in blockers calcium channels and with renal impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | Postoperative time while in hospital, up to 12 hours
  consumption of opioids and pain scores after surgery, during hospitalization.

SECONDARY OUTCOMES:
Magnesium blood concentration | At the time of venipuncture and 15, 30, 60, 120 and 240 minutes after the beginning of the covered solution.
  Blood will be collected to examine the blood concentration of magnesium in all patients in the 3 groups
Neuromuscular block recovery index | Intraoperative time
  Cisatracurium latency, cisatracurium duration 25, total duration of cisatracurium, cisatracurium recovery index

CONTACTS AND LOCATIONS:
Overall Officials: sebastião silva filho, Principal Investigator — Hospital da Sociedade de Beneficência Portuguesa d
Locations (2):
- Brazil (2):
  - Sebastião Ernesto Silva Filho, São José dos Campos, São Paulo
  - Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowther CA, Hiller JE, Doyle LW, Haslam RR; Australasian Collaborative Trial of Magnesium Sulphate (ACTOMg SO4) Collaborative Group. Effect of magnesium sulfate given for neuroprotection before preterm birth: a randomized controlled trial. JAMA. 2003 Nov 26;290(20):2669-76. doi: 10.1001/jama.290.20.2669. PMID 14645308
- [Background] Duley L, Meher S, Jones L. Drugs for treatment of very high blood pressure during pregnancy. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD001449. doi: 10.1002/14651858.CD001449.pub3. PMID 23900968
- [Background] Lu JF, Nightingale CH. Magnesium sulfate in eclampsia and pre-eclampsia: pharmacokinetic principles. Clin Pharmacokinet. 2000 Apr;38(4):305-14. doi: 10.2165/00003088-200038040-00002. PMID 10803454
- [Background] Jee D, Lee D, Yun S, Lee C. Magnesium sulphate attenuates arterial pressure increase during laparoscopic cholecystectomy. Br J Anaesth. 2009 Oct;103(4):484-9. doi: 10.1093/bja/aep196. Epub 2009 Jul 17. PMID 19617379
- [Background] James MF, Beer RE, Esser JD. Intravenous magnesium sulfate inhibits catecholamine release associated with tracheal intubation. Anesth Analg. 1989 Jun;68(6):772-6. PMID 2735543
- [Derived] S E SF, G F M, S D, M A M C G, F A, C B, F B S, J E V. Optimal Dose of Magnesium Sulfate Infusion in Obese Patients: A Double-Blind Randomized Trial. Anesthesiol Res Pract. 2025 Mar 19;2025:8854830. doi: 10.1155/anrp/8854830. eCollection 2025. PMID 40144953